CLINICAL TRIAL: NCT03757338
Title: A Randomized, Single Dose, Crossover, Bioequivalence Study of Fingolimod 0.5 mg Capsule (Asofarma S.A.I. y C., Argentina) Compared With Gilenya 0.5 mg Capsule (Novartis Pharmaceuticals, Australia Pty Ltd) in Fasting Healthy Subjects
Brief Title: Bioequivalence Study of a Test Capsule Formulation of Fingolimod With the Reference Capsule Formulation of Fingolimod
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asofarma S.A.I. y C. (Industry)
Collaborators: Zenith Technology Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ACTRN12615001055594; ZPS-578 (C15-020-LBB) (Registry Identifier: Zenith Code)
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single centre, single dose, blinded, two treatment, two period, two sequence, two-way crossover, randomized study.
Who Masked: Outcomes Assessor
Masking Description: The study was conducted as a blinded study regarding dose administration and sample collection. In addition, the blood samples from each subject were coded in a manner to make the analyst blind to the identity of the samples, allowing efficient conduct of the analytical procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fingolimod Reference Formulation (Active Comparator): 0.5 mg Fingolimod capsule (manufactured by Novartis, Batch No. S0099), orally administered as a single dose of 3 x 0.5 mg capsules.
  Interventions: Drug: Fingolimod Reference Formulation
- Fingolimod Test Formulation (Experimental): 0.5 mg Fingolimod capsule (manufactured by manufactured by Asofarma S.A.I. y C. on behalf of Tolmar, Batch No. 22264), orally administered as a single dose of 3 x 0.5 mg capsules.
  Interventions: Drug: Fingolimod Test Formulation

INTERVENTIONS:
Drug: Fingolimod Reference Formulation — To compare the rate and extent of absorption for Fingolimod when administered as a single oral dose of 3 x 0.5 mg capsules of the reference product produced by Novartis Pharmaceutical with the proposed test product manufactured by Asofarma S.A.I. y C. in healthy volunteers, under fasted conditions.
  Other Names: Gylenia®
  Arms: Fingolimod Reference Formulation
Drug: Fingolimod Test Formulation — To compare the rate and extent of absorption for Fingolimod when administered as a single oral dose of 3 x 0.5 mg capsules of the proposed test product manufactured by Asofarma S.A.I. y C. with the reference product produced by Novartis Pharmaceutical in healthy volunteers, under fasted conditions.
  Other Names: Lebrina®
  Arms: Fingolimod Test Formulation

SUMMARY:
The study evaluates the bioequivalence of the Test formulation, 0.5 mg Fingolimod HCl capsule (Asofarma S.A.I. y C. on behalf of Tolmar, Batch No. 22264), relative to that of the Reference formulation, 0.5 mg Gilenya® (fingolimod) capsule (Novartis Pharmaceuticals, Batch No. S0099), following oral administration of a single oral dose of 3 x 0.5 mg in healthy, adult, male and female subjects under fasting conditions.

DETAILED DESCRIPTION:
This was a single centre, single dose, blinded, two treatment, two period, two sequence, two-way crossover, randomized study conducted under medical supervision at Zenith Technology Corporation Limited's Clinical Site and involving 32 healthy adult subjects.

All subjects received either the Test or the Reference product under fasting conditions in each of the two treatment periods. In Period 1, one half of the subjects (16) were scheduled to receive 3 x 0.5 mg Fingolimod HCl capsules (Test); and one half of the subjects (16) were scheduled to receive 3 x 0.5 mg Gilenya® capsules (Reference). Each subject was scheduled to receive the alternate treatment in Period 2.

The two treatments were administered with 240 ml of ambient-temperature water after an overnight fast of at least 10 hours. Subjects did not receive any food until at least 4 hours post-dose. The capsules were swallowed whole.

During each study period, subjects were confined to the Zenith Clinical Site from at least 12 hours prior to drug administration, until after the 24-hour post-dose blood draw. Blood samples (18 x 10 ml) were collected at specified intervals during the in-house period from pre-dose (0 hours) out to 24 hours post-dose. Subjects returned to Zenith premises for the collection of additional blood samples (4 x 10 ml) at 32, 48, 56 and 72 hours post-dose. A total of 22 x 10 ml blood samples were collected in each study period.

The doses in the two treatment periods were separated by a washout period of at least 42 days and the project duration was 46 days for subject dosing and blood sampling over two periods.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for the participation in the study.
* Aged between 18 and 45 years, inclusive.
* All females of childbearing potential must have a negative serum pregnancy test 3 days prior to dosing in both study periods.
* Females of childbearing potential must agree to acceptable method of contraception (as agreed with the study doctor) or abstain from sexual activity during the study.
* Body Mass Index (BMI) within 18 - 30 kg/m2, inclusive, with body mass above 45 kg.
* Normal, healthy individuals as determined by medical history, physical examination, vital signs, ECG and laboratory tests.
* Non-smoker (for at least 6 months). This includes all tobacco products and nicotine containing patches and gums.
* Must abstain from consuming alcohol and caffeine and remain chocolate free for 48 hours prior to the study and throughout each study period (i.e. until 72 hours post-dosing in each period).
* Non-consumption of grapefruits or oranges, grapefruit and/or orange juice and any grapefruit and/or orange products for 1 week prior to the study and throughout the study (i.e. until 72 hours after receiving the final dose).
* Subjects must agree and be able to follow the study procedures, in the Investigator's opinion.

Exclusion Criteria:

* Known hypersensitivity to fingolimod, its analogues or excipients of the tested drug or the reference drug, lactose malabsorption, glucose-galactose malabsorption or Lapp lactase deficiency.
* Aggravated history of allergies (evidence of anaphylactic shock or Quincke's edema).
* History of gastrointestinal (GI), hepatic or renal abnormality or any other abnormality, which, in the Investigator's opinion, may affect absorption, distribution, metabolism and excretion of the IMPs (e.g. operative interventions to the GI tract other than appendectomy).
* Pregnant or breastfeeding females.
* Acute infectious diseases within 4 weeks before the study start.
* Significant cardio-vascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic, ophthalmologic or dermatologic disease.
* Subjects who have had any severe eye problems or conditions especially inflammation of the eye, such as uveitis.
* Vital signs measured in the seated position: heart rate <50 or >90 beats per minute or systolic BP <90 mmHg or >160 mmHg or diastolic BP <50 mmHg or >90 mmHg.
* Subjects with prolonged QTc interval (defined as >450 msec for males and >470 msec for females).
* Any clinically significant laboratory abnormalities at screening, including potassium, bilirubin, asparte transaminase (AST) and alanine transaminase (ALT) blood levels.
* Evidence of routine consumption of more than 10 units of alcohol per week within 6 months before screening (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of wine or 50 ml of spirit), positive breath test for alcohol or alcohol consumption within 48 hours prior to the study start.
* Evidence of any drug abuse within one year prior to the study start or positive urine drug and prohibited medication screen.
* Concomitant drug therapy of any kind with the exception of prescribed hormonal contraceptives.
* Having received vaccinations within 1 month prior to dosing or any planned vaccination within 2 months of the last dose of fingolimod.
* Administration of any medication that can cause a significant effect onto hemodynamics or liver function within 30 days prior to the study start.
* Administration of any medications which can induce or inhibit the drug hepatic metabolism via CYP1A2, CYP2D6, CYP2C8, CYP3A4 and CYP17 (hepatic metabolism inducers include barbiturates, carbamazepine, phenytoin, glucocorticosteroids, omeprazole; hepatic metabolism inhibitors include antidepressants, cimetidine, diltiazem, macrolides, imidazole, neuroleptics, verapamil, fluoroquinolones, antihistamine drugs), as well as herbal preparations and extracts within 30 days prior to the study start.
* Administration of any injectable deposit (sustained release) formulations or drug implants within 3 months prior to the study drug administration.
* Participation in any clinical study within 60 days prior to the study start.
* Donation or loss of more than 450 ml of blood within 2 months prior to the screening visit.
* Possible difficulties with study drug swallowing.
* History of tuberculosis or participation in the tuberculosis control program.
* Herpes simplex or varicella zoster virus infection including cold sore, genital herpes, chickenpox or shingles.
* Human Immunodeficiency Virus (HIV) positive test, positive test for hepatitis B or C.
* Other acute or chronic medical or mental conditions, laboratory abnormalities which may increase risk associated with the study participation or with study drug administration or which may affect interpretation of the study results and, in the Investigator's opinion, make the subject non-eligible for participation in this study.
* Inability of the subject to follow the requirements of the study.
* Employees of the study Sponsor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

PRIMARY OUTCOMES:
Fingolimod plasma Cmax (maximum plasma concentration) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod plasma Cmax will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod AUC0-t (area under the plasma concentration-time curve from time of intake until the last quantifiable concentration) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod AUC0-t will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod AUC0-∞ (area under the plasma concentration-time curve from time of intake until infinity) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod AUC0-∞ will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.

SECONDARY OUTCOMES:
Fingolimod elimination t1/2 (elimination half-life), when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod t1/2 will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod Tmax (time to Cmax), when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Tmax will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.

OTHER OUTCOMES:
Fingolimod Phosphate plasma Cmax (maximum plasma concentration) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Phosphate plasma Cmax will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod Phosphate AUC0-t (area under the plasma concentration-time curve from time of intake until the last quantifiable concentration ) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Phosphate AUC0-t will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod Phosphate AUC0-∞ (area under the plasma concentration-time curve from time of intake until infinity ) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Phosphate AUC0-∞ will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod Phosphate elimination t1/2 (elimination half-life) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Phosphate elimination t1/2 will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.
Fingolimod Phosphate Tmax (time to Cmax) when administered as a single oral dose of 3 x 0.5 mg capsule of the test versus reference product. | Measurement within 72 hours post-dose.
  Fingolimod Phosphate Tmax will be calculated based on plasma Fingolimod concentrations within 1 hour pre-dose (time 0) and at 1, 2, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 20, 24, 32, 48, 56 and 72 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Noelyn A Hung, MB ChB, Principal Investigator — Zenith Technology Corporation Ltd, 156 Frederick Street, Dunedin, New Zealand
Locations (1):
- Zenith Clinical Site, Dunedin, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Food and Drug Administration, USA. Bioequivalence Recommendations for fingolimod, Aug 2011.
- [Background] Australian Product Information, Gilenya, 1 April 2015
- [Derived] Hung NA, Costa FG, Hung CT, Rosenberg ME. Bioequivalence Study of 2 Capsule Formulations of Fingolimod 0.5 mg Assessing Both Parent Drug and Active Metabolite in New Zealand Healthy Subjects (Truncated Design). Clin Pharmacol Drug Dev. 2020 Jul;9(5):610-620. doi: 10.1002/cpdd.813. Epub 2020 May 28. PMID 32468719